CLINICAL TRIAL: NCT02666326
Title: Accelerated Rule-Out of Acute Myocardial Infarction, Using Copeptin and High Sensitive Troponin T - the AROMI Trial
Brief Title: Accelerated Rule Out of Myocardial Infarction
Acronym: AROMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, Associate professor, MD, DmSc, PhD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AROMI-1
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Myocardial Infarction
Keywords: Acute Coronary Syndrome; Prehospital emergency care; Biological markers; Copeptin; Troponin; Rule-out; Point-of-Care systems; Infarction; Cardiovascular Diseases; Heart Diseases; Ischemia; Myocardial Ischemia; copeptins; Troponin T; Diagnostic Techniques (Cardiovascular); High sensitivity troponin
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Diabetes Insipidus; Infarction; Cardiovascular Diseases; Heart Diseases; Ischemia; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional diagnostic strategy (No Intervention): Standard Diagnostics for suspected myocardial infarction, including standard biochemical analysis: min. two measurements of high sensitive troponin T with an interval of minimum 3 hours.
  A normal value of high sensitive cardiac troponin-T in both blood samples rules out AMI and the patients can be discharged immediately if no other conditions are suspected.
- Accelerated diagnostic strategy (Experimental): 'Accelerated, combined biomarker rule-out strategy for MI'. Copeptin measurement in a prehospital blood sample combined with high sensitive cardiac troponin T measurement in the first blood sample upon hospital admission, A normal value of both copeptin and cardiac troponin rules out AMI and the patients can be discharged immediately if no other conditions are suspected.
  Interventions: Procedure: Accelerated, combined biomarker rule-out strategy for MI

INTERVENTIONS:
Procedure: Accelerated, combined biomarker rule-out strategy for MI — Blood sample is acquired while the patient is in the ambulance. This is brought to hospital and handed over to the laboratory personnel for acute analysis for copeptin level. At arrival to hospital, a second blood sample is acquired and analyzed for high-sensitive cardiac troponin-T(hs-cTnT). Answers of these analyzes are in-hand with-in 60 minutes. If copeptin in the pre-hospital blood sample is <9,8 pmol/L (95% percentile) AND hs-cTnT in the in-hospital blood sample is <14ng/L (99% percentile), then myocardial infarction can be ruled out, and depending of clinical presentation, the patient can be discharged.
  Arms: Accelerated diagnostic strategy

SUMMARY:
Every year > 50.000 people in Denmark are hospitalized with a suspected acute myocardial infarction (AMI). The majority has other explanations of their chest discomfort and most are discharged again without any initiation of treatment. Still, the suspicion dictates acute ambulance deployment, hospital admission to a highly specialized cardiac unit, cardiac surveillance and cardiac troponin blood sampling. The novel biomarker copeptin, a byproduct of vasopressin production, is released immediately from the pituitary gland as part of the hormonal response to AMI. Peak concentrations are reached within the first hour. Previous studies have suggested the combination of copeptin and cardiac troponin for fast and reliable rule out of AMI. However, the blood sampling should be performed as soon as possible after symptom onset, preferably already during the prehospital phase.

We aim, in an open randomized setting, to investigate the combined measurement of prehospital copeptin and in-hospital high sensitive cardiac Troponin T compared to the standard rule-out procedure of suspected myocardial infarction. We hypothesize that the combined measurement of prehospital copeptin and in-hospital high sensitive troponin T:

1. Reduces admission time by 1.5 hours in patients where AMI is ruled out
2. Reduces the time to disposition
3. Is non-inferior compared to the standard rule-out procedure in relation to major adverse cardiovascular events.
4. Is more cost efficient compared to standard diagnostic strategy

DETAILED DESCRIPTION:
Patients with suspected Acute Myocardial Infarction (AMI) constitute one of the largest patient groups in emergency medicine. The majority of these patients, however, have other causes than AMI, for their chest discomfort and many are discharged again without any initiation of treatment.(1) At present, cardiac troponin is gold standard in diagnosing AMI. Diagnostic levels of troponin are not reached until hours after onset of symptoms and serial sampling is recommended at intervals of 3-6 hours to confirm or rule-out AMI. The novel biomarker copeptin, a by-product of vasopressin production, is released immediately from the pituitary gland as part of the hormonal response to AMI. However, copeptin elevation, is not specific of AMI. Peak concentrations of copeptin are reached within the first hour and the values normalizes within 4-10 hours.(3) Previous studies have suggested the combination of copeptin and high-sensitive cardiac troponin T (hs-cTnT) for early and reliable rule-out of AMI.(2,3,6) These studies are based on copeptin measurement in blood sample acquired at hospital admission. However, because of the rapid release of copeptin, the blood sampling should be performed as early as possible after symptom onset, preferably already in the ambulance, whereas the analysis can be performed after arrival at the hospital because copeptin is stable. The PREHAB trial conducted in the Central Denmark Region, documented that prehospital blood sampling is performed 70 minutes earlier than first in-hospital sample.(5) Post-trial analysis of blood samples from the PREHAP trial has demonstrated the potential for early and safe rule-out of AMI using the combination of prehospital copeptin and in-hospital troponin analysis. AMI could potentially be safely, ruled out in approximately 40-50% of patients, in whom the AMI diagnosis eventually was dismissed.

During the last 7 years, studies have evaluated the effect and validity of prehospital blood sample analysis. This is now standard procedure in The Central Denmark Region, Denmark.(5) Currently, prehospital blood sampling is carried out in two major randomized studies, aiming at identifying patients with myocardial infarction and heart failure (NCT01638806 and NCT02050282).

Unfortunately, there is at present no point-of-care analysis equipment for copeptin available. Manufacturer of copeptin analysis equipment, Thermo Fischer, has informed that the development of point-care-care equipment is in process, but will not be available in near future. Therefore, we will perform in-hospital analysis of the prehospital blood samples.

Overall aim of this protocol is to demonstrate the combination of troponin T and copeptin as a safe and effective biomarker for rule-out of AMI. In a randomized setting, we will compare the combination of prehospital copeptin and in hospital hs-cTnT, to the standard diagnostic procedure in patients with suspected AMI, evaluating rule-out potential and potential for reduction of the length of stay at the hospital. The diagnostic effects of measuring copeptin/ hs-cTnT in prehospital vs in-hospital blood samples will be evaluated. Moreover an other diagnostic rule-out strategy, using hs-cTNT at admission and 1 hour after admission, will be evaluated in retrospective analysis of blood samples acquired from patients in the conventional diagnostics arm of the study.

Primary purposes of the AROMI trial:

1. To evaluate if early discharge, based in the combined biomarker analysis is associated to duration of hospital stay. Will be evaluated in interim analysis after rule out of AMI(discharged within 12 hours) in 900 patients (300 patients in each site)
2. To evaluate if early discharge, based in the combined biomarker analysis is associated to major adverse cardiac events (MACE) during index admission, after discharge, within 30, 90, and 365 days of randomization (separately or in combination). No interim evaluation of MACE.

Secondary purposes of the AROMI trial:

1. To evaluate if early discharge, based in the combined biomarker analysis is associated to time to decision of discharge or continued hospitalization. Will be evaluated in interim analysis after rule out of AMI(discharged within 12 hours) in 900 patients (300 patients in each site)
2. To evaluate if early discharge, based in the combined biomarker analysis is cost-effective regarding satisfaction and safety from a patients perspective.
3. To evaluate if early discharge, based in the combined biomarker analysis is cost-effective from a public perspective, regarding staff resources, costs of hospital stay, adherence to the labour market, and use of other healthcare services, Cost benefit analysis(CBA).
4. To evaluate if early discharge, based on the hs-cTnT analysis at arrival and 1 hour after arrival at hospital is associated to duration of hospital stay.
5. To evaluate if early discharge, based on the hs-cTnT analysis at arrival and 1 hour after arrival at hospital is associated to MACE(major adverse cardiac event) during index admission, after discharge, within 30, 90, and 365 days of randomization (separately or in combination).
6. To evaluate the diagnostic properties (including sensitivity, specificity, negative predictive value, and positive predictive value) of the accelerated rule out algorithm using copeptin and high sensitivity troponin. Will be evaluated in interim analysis after rule out of AMI(discharged within 12 hours) in 900 patients (300 patients in each site). Will be evaluated in the total cohort (since both prehospital and inhospital copeptin and high sensitivity troponin is available in all patients) and randomization will not be revealed during this evaluation.
7. To evaluate the prognostic value of the accelerated rule out algorithm using copeptin and high sensitivity troponin. Will be evaluated in interim analysis after rule out of AMI(discharged within 12 hours) in 900 patients (300 patients in each site). Will be evaluated in the total cohort (since both prehospital and inhospital copeptin and high sensitivity troponin is available in all patients) and randomization will not be revealed during this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients which, after telemedical triage, are admitted to a cardiac department in suspicions of myocardial infarction
* A peripheral venous catheter has been inserted prehospitally and blood has drawn from it, before flushing it.

Exclusion Criteria:

* Age below 18 years
* Patients in which an informed concent can not be obtained (psychiatric disease, dementia, under influence of drugs etc.),
* Suspected STEMI and referral to Primary percutaneous coronary intervention (PPCI), referral to a highly specialized cardiac department for another cardiac reason (e.g ventricular tachycardia, ventricular fibrillation, 3° Atrio-ventricular block.)
* Known central Diabetes insipidus
* Other diagnosis as obvious reason for symptoms at time of admittance (e.g. a new diagnosis of supraventricular tachycardia, pulmonary embolism, aortic dissection) AND no suspicions of ACS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4516 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | Up to three months from randomization
  Time (hours and minutes) from admission to discharge from cardiac department. Reported by clinical personnel in registration form and supplemented by data from the national health registry. Will be evaluated in interim analysis after inclusion of 300 patients in each site.
Combined MACE | Within time from randomization to 30 days after randomization
  Combined endpoint of major adverse cardiac events, consisting of: "All-cause mortality", "survived cardiac arrest", "Confirmed or Readmission with Acute Coronary Syndrome(ACS)", "Non-scheduled coronary intervention", and "Life-threatening arrhythmias" (see below for description) occuring within time from randomization to 30 days after randomization

SECONDARY OUTCOMES:
Time to disposition | Within 24 h of randomization
  Time from admission to decision of early discharge or continued admission for further diagnostics or treatment. Will be evaluated in interim analysis after inclusion of 300 patients in each site.
Combined MACE | Within index admission, within time from discharge to 30, 90, and 365 days after randomization, and within time from randomization to 90 and 365 days after randomization
  Combined endpoint of major adverse cardiac events, consisting of: "All-cause mortality", "survived cardiac arrest", "Readmission with Acute Coronary Syndrome(ACS)", "Non-scheduled coronary intervention", and "Life-threatening arrhythmias" (see below for description)
All-cause mortality | Within index admission and within 30, 90 and 365 days of randomization
  All-cause mortality registered in the national health registry, occurring from time of admission to discharge, within 30, 90 or 365 days after randomization.
Survived, cardiac arrest | Within index admission and within 30, 90 and 365 days of randomization
  Survived cardiac arrest is determined from registration of out-of-hospital cardiac arrest in "Danish register of cardiac arrest" or in-hospital cardiac arrest in "Danarrest" or in the national health registry, occurring from time of admission to discharge, within 30, 90 or 365 days after randomization. The endpoint committee adjudicate survived cardiac arrest, blinded to the initial randomization.
Confirmed diagnosis of ACS or readmission with ACS | Within index admission and within 30, 90 and 365 days of randomization
  The national health registry is used to determine whether the patient is confirmed of having or readmitted with acute coronary syndrome, from time of admission to discharge and within 30, 90 or 365 days after randomization. The endpoint committee adjudicate readmission with acute coronary syndrome, blinded to the initial randomization. The "2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation" and "Universal definition of Myocardial infarction" will be used to evaluate if the patient had: ACS, and subsequently classify it as a: a) Unstable angina pectoris(UAP), b) non-ST-elevation myocardial infarction (NONSTEMI), c) ST-Elevation myocardial infarction (STEMI) d) Bundle branch block myocardial infarction (BBBMI)
Non-scheduled coronary intervention | Within index admission and within 30, 90 and 365 days of randomization
  The national health registry is used to determine whether the patient has non-scheduled re-intervention performed (re-intervention not scheduled at index admission). Time from index admission to first re-intervention and type of re-intervention (PCI or CABG) is determined. The endpoint committee adjudicate re-interventions blinded to original treatment strategy
Life-threatening arrhythmias | Within index admission and within 30, 90 and 365 days of randomization
  The national health registry is used to determine whether the patient is diagnosed or readmitted with a life-threatening arrhythmia, defined as ventricular tachycardia, ventricular fibrillation or third-degree(total) atrioventricular block within index admission and within 30, 90 or 365 days of randomization. The endpoint committee adjudicate readmission with life-threatening arrhythmia, blinded to the initial randomization.

OTHER OUTCOMES:
Cost efficiency | Within index admission, and 1 year after randomization
  Costs and cost effectiveness will be evaluated and compared between the two diagnostic strategies.
Risk factors and patient experiences | Within index admission, and 1 year after randomization
  The patients experience of being discharged earlier and risk factors for early readmission.
Myocardial injury | Within index admission
  The laboratory registries is used to determine whether the patient has troponin elevation, from time of admission to discharge. The endpoint committee adjudicate myocardial injury, blinded to the initial randomization. "Universal definition of Myocardial infarction" will be used to evaluate the event.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Stengaard, MD, PhD, Study Chair — Aarhus University Hospital Skejby; Hanne M Soendergaard, MD, PhD, Study Chair — Viborg Regional Hospital; Christian J Terkelsen, MD, DmSc, Associate prof., Study Chair — Aarhus University Hospital Skejby; Karen K Dodt, MD, PhD, Study Chair — Regionshospitalet Horsens
Locations (3):
- Denmark (3):
  - Department of Cardiology, Viborg Regional Hospital, Viborg, Central Jutland
  - Department of Cardiology, Aarhus University Hospital, Aarhus
  - Department of Internal Medicine, Horsens Regional Hospital, Horsens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grande P, H. L. Akut koronar syndrom, retningslinier for diagnostik og behandling. Dansk Cardiologisk Selskab. 2004 Download from http://www.cardio.dk/docman/doc_download/149-akut-koronart-syndrom. (danish)
- [Background] Maisel A, Mueller C, Neath SX, Christenson RH, Morgenthaler NG, McCord J, Nowak RM, Vilke G, Daniels LB, Hollander JE, Apple FS, Cannon C, Nagurney JT, Schreiber D, deFilippi C, Hogan C, Diercks DB, Stein JC, Headden G, Limkakeng AT Jr, Anand I, Wu AHB, Papassotiriou J, Hartmann O, Ebmeyer S, Clopton P, Jaffe AS, Peacock WF. Copeptin helps in the early detection of patients with acute myocardial infarction: primary results of the CHOPIN trial (Copeptin Helps in the early detection Of Patients with acute myocardial INfarction). J Am Coll Cardiol. 2013 Jul 9;62(2):150-160. doi: 10.1016/j.jacc.2013.04.011. Epub 2013 Apr 30. PMID 23643595
- [Background] Morgenthaler NG. Copeptin: a biomarker of cardiovascular and renal function. Congest Heart Fail. 2010 Jul;16 Suppl 1:S37-44. doi: 10.1111/j.1751-7133.2010.00177.x. PMID 20653710
- [Background] Reinstadler SJ, Klug G, Feistritzer HJ, Metzler B, Mair J. Copeptin testing in acute myocardial infarction: ready for routine use? Dis Markers. 2015;2015:614145. doi: 10.1155/2015/614145. Epub 2015 Apr 16. PMID 25960596
- [Background] Stengaard C, Sorensen JT, Ladefoged SA, Christensen EF, Lassen JF, Botker HE, Terkelsen CJ, Thygesen K. Quantitative point-of-care troponin T measurement for diagnosis and prognosis in patients with a suspected acute myocardial infarction. Am J Cardiol. 2013 Nov 1;112(9):1361-6. doi: 10.1016/j.amjcard.2013.06.026. Epub 2013 Aug 14. PMID 23953697
- [Background] Mockel M, Searle J, Hamm C, Slagman A, Blankenberg S, Huber K, Katus H, Liebetrau C, Muller C, Muller R, Peitsmeyer P, von Recum J, Tajsic M, Vollert JO, Giannitsis E. Early discharge using single cardiac troponin and copeptin testing in patients with suspected acute coronary syndrome (ACS): a randomized, controlled clinical process study. Eur Heart J. 2015 Feb 7;36(6):369-76. doi: 10.1093/eurheartj/ehu178. Epub 2014 Apr 30. PMID 24786301
- [Derived] Pedersen CK, Stengaard C, Botker MT, Sondergaard HM, Dodt KK, Terkelsen CJ. Accelerated -Rule-Out of acute Myocardial Infarction using prehospital copeptin and in-hospital troponin: The AROMI study. Eur Heart J. 2023 Oct 12;44(38):3875-3888. doi: 10.1093/eurheartj/ehad447. PMID 37477353
- [Derived] Pedersen CK, Stengaard C, Sondergaard H, Dodt KK, Hjort J, Botker MT, Terkelsen CJ. A multicentre, randomized, controlled open-label trial to compare an Accelerated Rule-Out protocol using combined prehospital copeptin and in-hospital high sensitive troponin with standard rule-out in patients suspected of acute Myocardial Infarction - the AROMI trial. Trials. 2018 Dec 12;19(1):683. doi: 10.1186/s13063-018-2990-z. PMID 30541594